CLINICAL TRIAL: NCT00774358
Title: Reinstituting Natural Killer Cell Cytotoxicity and Cytoskeletal Dynamics in Wiskott-Aldrich Syndrome With IL-2 Therapy
Brief Title: Interleukin-2 Treatment for Wiskott-Aldrich Syndrome
Acronym: WAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soma Jyonouchi (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Soma Jyonouchi, Soma Jyonouchi,MD, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-6-5354; 1R01FD004091-01A1 (FDA)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2016-09

CONDITIONS: Wiskott-Aldrich Syndrome (WAS); X-linked Thrombocytopenia
Keywords: Primary Immunodeficiency
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Thrombocytopenia 1; Primary Immunodeficiency Diseases | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 (Experimental): We propose to subcutaneously administer 0.5 MU/m2 of IL-2 daily to WAS subjects for 5 days. Research treatment will be repeated 2 and 4 months later. Inter-patient dose escalation will be employed to 1 MU/m2 and/or 2 MU/m2 based on safety as the primary endpoint.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — We propose to subcutaneously administer 0.5 MU/m2 of IL-2 daily to WAS subjects for 5 days. Research treatment will be repeated 2 and 4 months later. Inter-patient dose escalation will be employed to 1 MU/m2 and/or 2 MU/m2 based on safety as the primary endpoint.
  Other Names: IL-2; Aldesleukin; Proleukin

SUMMARY:
Funding Source--FDA OOPD.

Orphan Product Grant Number--1R01FD004091-01A1

Context: Wiskott-Aldrich syndrome (WAS) is a fatal, devastating disease with ill-defined treatment modalities, which affects young boys. Classic WAS is characterized by a clinical triad of thrombocytopenia, eczema and severe, recurrent infections. Despite diagnostic and therapeutic advances most WAS patients die at less than 12 years of age due to infections, hemorrhage, malignancy or complications from treatments. WAS patients suffer from herpesvirus infections as a result of poor Natural Killer (NK) cell function (cytotoxicity). In the laboratory, the investigators have seen correction of WAS Natural Killer Cell (NK) function after treatment with Interleukin-2 (IL-2).

Objectives: Initiate a prospective clinical trial by treating WAS subjects with IL-2 and using safety as the primary endpoint. Restoration of NK cell cytotoxicity and effects on cytoskeletal dynamics are secondary endpoints. The investigators will also observe patient clinical status (eczema, infections, use of treatment dose antibiotics, food allergies, etc).

Study Design/Setting/Participants: This is a prospective clinical trial treating 9 WAS subjects in the Clinical Translational Research Center (CTRC) with IL-2.

Intervention: The investigators propose to subcutaneously administer 0.5 Million Units (MU)/m2 of IL-2 daily to WAS subjects for 5 days. Research treatment will be repeated 2 and 4 months later. Inter-patient dose escalation will be employed to 1 MU/m2 and/or 2 MU/m2 based on safety as the primary endpoint.

Study Measures: The investigators will observe safety and tolerability measures and perform assays on subject blood samples prior to and after research treatment to observe improvement in NK cell function.

DETAILED DESCRIPTION:
The Wiskott-Aldrich syndrome (WAS) is a fatal genetic disease of the immune system that results from a mutation of the WAS protein (WASp) gene. Immune cells that carry this mutation have a decreased ability to reorganize filamentous actin (F-actin) after activation. As a result there are a number of defective immunologic functions, some of which result in deficient host defense. The investigators have identified a pervasive deficit in natural killer (NK) cell cytotoxicity in WAS patients. WAS patients suffer from conditions that are hallmarks of NK cell deficiencies. These include severe herpesvirus infections and B cell malignancies. Our lab and others have also found that exposure of WAS subject NK cells to IL-2 in vitro restores NK cell function and allows for normal F-actin reorganization. Thus, the investigators propose a proof of principal clinical trial to treat WAS subjects with IL-2 to determine safety and efficacy of IL-2 in this population and if NK cell function is restored ex vivo. If IL-2 can circumvent a defective WASp to restore NK cell function, the investigators will propose a larger NIH funded efficacy trial of IL-2 in WAS. The investigators will also use the in vivo treatment of WAS subjects to forward our mechanistic studies of how IL-2 may facilitate F-actin reorganization in the absence of WASp function.

ELIGIBILITY:
Inclusion Criteria:

* Age: Subjects age greater than 24 months
* Weight: Subjects greater than 12.5 kilograms
* Disease status: WAS classified as Grade 1-4
* Informed Consent: Written informed consent of the subject (if an adult) or parental permission, and assent of the child subject provided justification is made for the inclusion of children in the study

Exclusion Criteria:

* Prior or planned hematopoetic transplant
* WAS classified as currently Grade 5 (Malignancy or autoimmune disease including the following: Crohn's disease, scleroderma, thyroiditis, inflammatory arthritis, diabetes mellitus, oculo-bulbar myasthenia gravis, crescentic IgA glomerulonephritis, cholecystitis, cerebral vasculitis, Stevens-Johnson syndrome and bullous pemphigoid . Not included here are: Hepatitis C virus induced vasculitis, alopecia areata and systemic lupus erythematosus.)
* Known previous reaction to IL-2
* Subjects taking immunosuppressive medications that might alter study results
* Subjects taking nephrotoxic, cytotoxic, cardiotoxic, or hepatotoxic medications (including medications for hypertension)
* Subjects currently taking systemic corticosteroids (not included here: topical and inhaled corticosteroids)
* Subjects taking Interferon alpha
* Use of any other investigational agent in the last 30 days
* Women of childbearing potential not using contraception method(s), as well as women who are breastfeeding
* Subjects with abnormal cardiac, hepatic and CNS function

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 1 year

SECONDARY OUTCOMES:
Evaluate effects on cytoskeletal dynamics | 1 year
Requirement for treatment dose antibiotics | 1 year
Number and severity of infections | 1 year
Eczema | 1 year
Food allergies | 1 year
NK cell cytotoxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Soma Jyonouchi, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Azuma H, Sakata H, Saijyou M, Okuno A. Effect of interleukin 2 on intractable herpes virus infection and chronic eczematoid dermatitis in a patient with Wiskott-Aldrich syndrome. Eur J Pediatr. 1993 Dec;152(12):998-1000. doi: 10.1007/BF01957224. PMID 8131820
- [Background] Pahwa R, Chatila T, Pahwa S, Paradise C, Day NK, Geha R, Schwartz SA, Slade H, Oyaizu N, Good RA. Recombinant interleukin 2 therapy in severe combined immunodeficiency disease. Proc Natl Acad Sci U S A. 1989 Jul;86(13):5069-73. doi: 10.1073/pnas.86.13.5069. PMID 2787027
- [Background] Piscitelli SC, Wells MJ, Metcalf JA, Baseler M, Stevens R, Davey RT Jr. Pharmacokinetics and pharmacodynamics of subcutaneous interleukin-2 in HIV-infected patients. Pharmacotherapy. 1996 Sep-Oct;16(5):754-9. PMID 8888071
- [Background] Witzke O, Winterhagen T, Reinhardt W, Heemann U, Grosse-Wilde H, Kreuzfelder E, Roggendorf M, Philipp T. Comparison between subcutaneous and intravenous interleukin-2 treatment in HIV disease. J Intern Med. 1998 Sep;244(3):235-40. doi: 10.1046/j.1365-2796.1998.00365.x. PMID 9747746
- [Background] Toren A, Nagler A, Rozenfeld-Granot G, Levanon M, Davidson J, Bielorai B, Kaplinsky C, Meitar D, Mandel M, Ackerstein A, Ballin A, Attias D, Biniaminov M, Rosenthal E, Brok-Simoni F, Rechavi G, Kaufmann Y. Amplification of immunological functions by subcutaneous injection of intermediate-high dose interleukin-2 for 2 years after autologous stem cell transplantation in children with stage IV neuroblastoma. Transplantation. 2000 Oct 15;70(7):1100-4. doi: 10.1097/00007890-200010150-00019. PMID 11045650
- [Background] Sundin DJ, Wolin MJ. Toxicity management in patients receiving low-dose aldesleukin therapy. Ann Pharmacother. 1998 Dec;32(12):1344-52. doi: 10.1345/aph.18019. PMID 9876817
- [Background] Starr SE, McFarland EJ, Muresan P, Fenton T, Pitt J, Douglas SD, Deveikis A, Levin MJ, Rathore MH; PACTG 299 Study Team. Phase I/II trial of intravenous recombinant interleukin-2 in HIV-infected children. AIDS. 2003 Oct 17;17(15):2181-9. doi: 10.1097/00002030-200310170-00006. PMID 14523275
- [Background] Gismondi A, Cifaldi L, Mazza C, Giliani S, Parolini S, Morrone S, Jacobelli J, Bandiera E, Notarangelo L, Santoni A. Impaired natural and CD16-mediated NK cell cytotoxicity in patients with WAS and XLT: ability of IL-2 to correct NK cell functional defect. Blood. 2004 Jul 15;104(2):436-43. doi: 10.1182/blood-2003-07-2621. Epub 2004 Mar 4. PMID 15001467
- [Background] Orange JS, Brodeur SR, Jain A, Bonilla FA, Schneider LC, Kretschmer R, Nurko S, Rasmussen WL, Kohler JR, Gellis SE, Ferguson BM, Strominger JL, Zonana J, Ramesh N, Ballas ZK, Geha RS. Deficient natural killer cell cytotoxicity in patients with IKK-gamma/NEMO mutations. J Clin Invest. 2002 Jun;109(11):1501-9. doi: 10.1172/JCI14858. PMID 12045264
- See also: Please see Study Description at www.wastherapy.com — http://www.wastherapy.com